CLINICAL TRIAL: NCT02585622
Title: Novel Stromal Cell Therapy for Diabetic Kidney Disease (NEPHSTROM Study)
Brief Title: NEPHSTROM for Diabetic Kidney Disease
Acronym: NEPHSTROM
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: IMP NEPHSTROM ORBECEL-M is expired and additional extension is not feasible. Low recruitment rate at Birmingham center.
Sponsor: Mario Negri Institute for Pharmacological Research (Other)
Collaborators: Leiden University Medical Center (Other); Papa Giovanni XXIII Hospital (Other); Istituto Di Ricerche Farmacologiche Mario Negri (Other); Belfast Health and Social Care Trust (Other); National University of Ireland, Galway, Ireland (Other); University Hospital Birmingham, NHS Foundation Trust, Hospital, Birmingham, UK (Unknown); NHS Blood and Transplant (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: NEPHSTROM; 2016-000661-23 (EudraCT Number)
Record Dates: First submitted 2015-10-22; First posted 2015-10-23 (Estimated); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Diabetic Kidney Disease
Keywords: Diabetic Kidney Disease; Mesenchymal Stromal Cells (MSC); immune response; allogeneic; disease progression
MeSH Terms: conditions — Diabetic Nephropathies; Disease Progression

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bone marrow-derived Mesenchymal Stromal Cells (Experimental)
  Interventions: Biological: Mesenchymal Stromal Cells
- Cryostor CS10 (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Mesenchymal Stromal Cells — Cells will be administered intravenously at 3 different doses (80, 160, or 240 x 10^6, fixed dose) over 10-20 minutes. Volume total of fluid infused: 40 ml
  Other Names: Allogeneic Cellular Therapy (NEPHSTROM ORBCEL-M)
  Arms: Bone marrow-derived Mesenchymal Stromal Cells
Other: Placebo — Volume total of fluid infused: 40 ml
  Other Names: Cryostor CS10
  Arms: Cryostor CS10

SUMMARY:
The study will investigate, primarily, the safety, feasibility and tolerability and, secondarily, the preliminary efficacy of an allogeneic bone marrow-derived Mesenchymal Stromal Cell (MSC) therapy (ORBCEL-M) in study subjects with type 2 diabetes (T2D) and progressive diabetic kidney disease (DKD).

ELIGIBILITY:
Inclusion Criteria:

* Male and female ≥ 40 years and <85 years old. ;
* T2D for 3 or more years under a clinician with mandated responsibility for management of the patients to national guidelines;
* Urinary albumin excretion (UAE) ≥ 60 µg/min (in a 24 hour urine collection) and urine albumin-to-creatinine ratio (UACR) ≥ 88 mg/g (≥ 10 mg/mmol) (in a spot morning urine collection);
* Estimated GFR (eGFR) 30-50 ml/min/1.73 m^2 by the CKD-EPI equation on 2 or more consecutive measurements at least 30 days apart within the past 6 months;
* A documented decline of eGFR of ≥ -10ml/min/1.73 m^2 over the past 3 years or documented rate of eGFR decline of ≥ -5 ml/min/1.73 m^2 year based on 3 or more consecutive readings at least 90 days apart in the past 18 months;
* Lack of suspicion of renal diagnosis other than DKD;
* Willing and able to provide written informed consent.

Exclusion Criteria:

1. Current resting systolic BP ≥ 150 mmHg and current resting diastolic BP ≥ 90 mmHg in a clinical setting, despite treatment with 3 hypertensive agents of different classes (including one diuretic), measured in a quiet environment with morning medications already taken;
2. Initiation of a new anti-hypertensive agent within the past 6 months
3. Increase the dose of an anti-hypertensive agent by ≥ 100% of the previous dose within the past 3 months

   Exclusion criteria related to glycaemic control:
4. Current HbA1c > 75 mmol/mol (> 9%)
5. Initiation of a new hypoglycaemic agent within the past 6 months
6. Increase the dose of a hypoglycaemic agent by ≥ 100% of the previous dose within the past 3 months

   Exclusion criteria related to dyslipidaemia:
7. Current fasting total cholesterol > 7 mmol/l
8. Current fasting total triglycerides > 3.5 mmol/l
9. Initiation of a new lipid lowering agent within the past 6 months

   Other exclusion criteria:
10. Chronic lung or liver disease;
11. Cardiovascular events (myocardial infarction, stroke or acute limb ischemia) within 6 months prior to enrolment;
12. Current or history within 6 months prior to enrolment of NYHA class III or IV heart failure;
13. Other concomitant disease or conditions in the opinion of the investigator that are likely to pose risk to the patient and that would render the patient unsuitable for participation or that could impair patient safety or ability to participate in the study, such as active malignancy;
14. Irreversible disease or condition for which 6-month mortality is estimated to be greater than 50%;
15. Positive screening test for clinically significant anti-HLA antibodies. An initial antibody screening with Luminex® multi-antigen beads to detect class I and class II MHC antibodies followed by a Luminex single antigen bead assay to determine the specificity of any antibody detected. Potential study subjects with positive screening for any clinically significant anti-HLA antibody will be excluded and will not be eligible to participate in the NEPHSTROM clinical study (MFI>1500);
16. History or presence of any medical condition or disease which, in the opinion of the Investigator may place the participant at unacceptable risk for study participation;
17. Childbearing potential without use of effective acceptable methods of contraception. Women of childbearing potential can only be included in the study if a pregnancy test is negative at the screening visit (V1) and at baseline visit (V2) if they agree to use adequate contraception. Adequate contraception is defined as any combination of at least two effective methods of birth control, of which at least one is a physical barrier (e.g. condoms with hormonal contraception or implants or combined oral contraceptives, certain intrauterine devices). Women are considered post-menopausal and not of child-bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g. age appropriate) or 6 months of spontaneous amenorrhea with serum FSH levels > 40 mIU/mL or have had surgical treatment such as bilateral tubal ligation, bilateral oophorectomy, or hysterectomy.
18. Pregnancy or lactating;
19. Participation in other investigational medicinal product (IMP) trials within 30 days before the inclusion or concurrent to this study (18 month follow-up);
20. Inability to understand the potential risks and benefits of the study;
21. Legal incapacity.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2017-12-11 (Actual); Primary Completion 2022-11-03 (Actual); Study Completion 2024-01-03 (Actual)

PRIMARY OUTCOMES:
Number and severity of all pre-specified infusion-associated events and the overall number and frequency of adverse events. | Changes from baseline to study completion, up to 18 months after cell or placebo infusion.
  At each visit overall clinical condition of the patient will be evaluated and any adverse event wil be recorded.

SECONDARY OUTCOMES:
Glomerular filtration rate (GFR) | Changes from baseline up to 18 months after cell or placebo infusion.
  GFR will be measured by plasma clearance of unlabelled exogenous marker Iohexol and estimated by CKD-EPI and MDRD equations.
Urinary Albumin/Creatinine Ratio (ACR) | Changes from baseline at 6 months and then every six months to study completion,up to 18 months after cell or placebo infusion.
  ACR will be measured on spot morning urine samples.
Urinary albumin excretion (UAE). | Changes from baseline at 6 months and then every six months to study completion,up to 18 months after cell or placebo infusion.
  UAE will be measured on 24h urine samples using standardized methods.
Fasting blood glucose (target <126mg/dL) | Proportion of study participants within target range (<126mg/dL) at baseline and at each time point (day 1, day 7, month 1,3,6,12,18 after cell or placebo infusion).
HbA1c (target <75mmol/mol or <9%) | Proportion of study participants within target range (<75mmol/mol or <9%) at baseline and at each time point (day 1, day 7, month 1,3,6,12,18 after cell or placebo infusion).
Total cholesterol (target <200 mg/dl) | Proportion of study participants within target range (<200 mg/dl) at baseline and at each time point (day 1, day 7, month 1,3,6,12,18 after cell or placebo infusion).
LDL cholesterol (target <100 mg/dl) | Proportion of study participants within target range (<100 mg/dl) at baseline and at each time point (day 1, day 7, month 1,3,6,12,18 after cell or placebo infusion).
Triglycerides (target <170 mg/dl) | Proportion of study participants within target range (<170 mg/dl) at baseline and at each time point (day 1, day 7, month 1,3,6,12,18 after cell or placebo infusion).
Arterial blood pressure (the target value <130/80 mmHg) | Proportion of study participants within target range (<130/80 mmHg)at baseline and at each time point (day 1, day 7, month 1,3,6,12,18 after cell or placebo infusion).
Quality of life | Changes from baseline to 1,3,6,12 and 18 months after cell or placebo infusion.
  Quality of life will be evaluated by the administration of SF36 questionnaire.
Quality of life | Changes from baseline to 1,3,6,12 and 18 months after cell or placebo infusion.
  Quality of life will be evaluated by the administration of EQ-5D-5L questionnaire.
Anti-HLA antibody development | Changes from baseline to 3,12 and 18 months after cell or placebo infusion.
Inflammation and fibrosis related soluble mediators | Changes from baseline to 7 days, 1,6,12 and 18 months after cell or placebo infusion.
  Blood and urine bio-chip-based multiplex assay
Serum/plasma concentrations (pg/ml) of biomarkers of inflammation. | Changes from baseline to 7 days, 1,6,12 and 18 months after cell or placebo infusion.
  Biomarkers will include sTNFR1, sTNFR2, Il-6,TNF-alfa, IL-1beta, MCP-1 (CCL2), IL-8, FGF21.
Serum/plasma concentrations (ng/ml) of biomarkers of CKD progression. | Changes from baseline to 7 days, 1,6,12 and 18 months after cell or placebo infusion.
  Biomarkers will include Cystatin C, NGAL, Adiponectin, Leptin.
Urine concentrations (pg/ml adjusted to urine creatinine concentration) of biomarkers of inflammation. | Changes from baseline to 7 days, 1,6,12 and 18 months after cell or placebo infusion.
  Biomarkers will include sTNFR1, sTNFR2, Il-6,TNF-alfa, IL-1beta, MCP-1 (CCL2), IL-8.
Proportion/total number of circulating T cells, B cells, NK cells, monocytes, dendritic cells | Changes from baseline to 7 days, 1,6,12 and 18 months after cell or placebo infusion.
Cost-effectiveness of cell therapy | Changes from baseline to 1,3,6,12 and 18 months after cell or placebo infusion.
  Cost-effectiveness of cell therapy will be evaluated by providing the patients with a healthcare resource diary.

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Remuzzi, MD, Study Chair — ASST Papa Giovanni XXIII, Bergamo, Italy/IRCCS - Mario Negri Institute for Pharmacological Research; Mattew Griffin, MD, Principal Investigator — National University of ireland - Galway University Hospital -Regenerative Medicine Institute; Paul Cockwell, MD, Principal Investigator — University Hospital Birmingham NHS Foundation Trust; Peter Maxwell, MD, Principal Investigator — Belfast Health and Social Care Trust - Belfast City Hospital
Locations (4):
- National University of ireland - Galway University Hospital -Regenerative Medicine Institute, Galway, Ireland
- ASST - Papa Giovanni XXIII - U.O. Nefrologia e Dialisi/ Mario Negri Institute for Pharmacological Research - Clinical Research Center for Rare Diseases Aldo e Cele Daccò, Bergamo, BG, Italy
- United Kingdom (2):
  - Belfast Health and Social Care Trust - Belfast City Hospital, Belfast
  - University Hospital Birmingham NHS Foundation Trust - Queen Elizabeth Medical Centre, Birmingham

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Perico N, Remuzzi G, Griffin MD, Cockwell P, Maxwell AP, Casiraghi F, Rubis N, Peracchi T, Villa A, Todeschini M, Carrara F, Magee BA, Ruggenenti PL, Rota S, Cappelletti L, McInerney V, Griffin TP, Islam MN, Introna M, Pedrini O, Golay J, Finnerty AA, Smythe J, Fibbe WE, Elliman SJ, O'Brien T; NEPHSTROM Trial Consortium. Safety and Preliminary Efficacy of Mesenchymal Stromal Cell (ORBCEL-M) Therapy in Diabetic Kidney Disease: A Randomized Clinical Trial (NEPHSTROM). J Am Soc Nephrol. 2023 Oct 1;34(10):1733-1751. doi: 10.1681/ASN.0000000000000189. Epub 2023 Aug 10. PMID 37560967
- [Derived] Lu B, Lerman LO. MSC therapy for diabetic kidney disease and nephrotic syndrome. Nat Rev Nephrol. 2023 Dec;19(12):754-755. doi: 10.1038/s41581-023-00776-z. No abstract available. PMID 37783947